CLINICAL TRIAL: NCT05217004
Title: Systematic Evaluation of Mobile Applications for Informal Caregivers of People Living With Dementia
Brief Title: Evaluation of Mobile Apps for Informal Caregivers of People Living With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-177
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2022-02

CONDITIONS: Caregiver Burden; Stress; Dementia
Keywords: Apps; mhealth
MeSH Terms: conditions — Caregiver Burden; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dementia Talk (Experimental): Participants in this group will be asked to use the mobile app Dementia Talk over a 2-week period.
  Interventions: Other: Dementia Talk mobile application
- CLEAR Dementia Care (Experimental): Participants in this group will be asked to use the mobile app CLEAR Dementia Care over a 2-week period.
  Interventions: Other: CLEAR Dementia Care mobile application
- Waitlist Control Group (No Intervention): Participants in this group will not use any of the apps.

INTERVENTIONS:
Other: Dementia Talk mobile application — The app includes features for caregivers such as medication management, behavior symptom management and monitoring, stress management tips and strategies, and task management with other care providers.
  Arms: Dementia Talk
Other: CLEAR Dementia Care mobile application — The app provides information about dementia (e.g., types and symptoms of dementia) and allows caregivers to record, monitor, and chart behaviors in the care recipient.
  Arms: CLEAR Dementia Care

SUMMARY:
The purpose of this study is to evaluate the effectiveness of two currently available apps for unpaid caregivers of people living with dementia.

DETAILED DESCRIPTION:
Informal caregivers of people living with dementia experience stressors that are associated with adverse health outcomes. Mobile applications (i.e., apps) could potentially improve the delivery and increase access to interventions. Although apps for informal caregivers of people living with dementia are available, empirical evidence to support their effectiveness is limited. The evaluation will be conducted by recruiting informal caregivers of people living with dementia. Participants will be randomly assigned to one of the two app-using groups or a wait-list condition. In the rare event that a participant experiences issues downloading an assigned app (and before commencing the 2-week period), participants will be randomly assigned to one of the other two conditions. Participants in the app-using groups will be asked to use their app for a 2-week period, and burden, stress, overall health, and knowledge will be assessed before, after the 2-week period, and at a 3-week follow-up. Subjective app ratings and usability of apps will be collected after the 2-week period. A 3 between (group) by 3 within (time: baseline, post, follow-up) mixed model (repeated measures) multivariate analysis of variance and univariate analyses will be conducted to examine improvements on outcome measures over time. Interviews will be conducted, and textual data will be analyzed thematically to examine caregiver experiences, perceptions of caregivers in using selected apps, and preferences and needs of caregivers in the development of future apps. Findings from the proposed investigation can help guide caregivers in choosing the apps that best address their needs. Moreover, findings from the investigation can inform future developments of apps to address the needs of caregivers of people living with dementia.

ELIGIBILITY:
Inclusion Criteria:

* providing informal care for a person living with dementia (e.g., informal caregivers who are non-professionals; this may include immediate family members such as spouses, children, and other relatives, friends)
* living with or providing primary care for the person living with dementia (i.e., the care recipient is not in a long-term care facility)
* providing unpaid care
* own a smartphone (i.e., an iPhone or Android and/or can access either IOS or Android platforms)

Exclusion Criteria:

- using an app for caregiver stress/burden

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Zarit Caregiver Burden Interview (ZBI) total scores at 2 weeks | The ZBI will be administered at baseline (i.e., prior to starting the study) and immediately after the end of the intervention period (i.e., after a 2-week period).
  Caregiver burden will be assessed using the ZBI. The ZBI is a 22-item self-report questionnaire designed to measure the extent of the burden experienced by the caregivers in various dimensions (e.g., health, psychological well-being, finances, social) of their lives as a result of caregiving. Each item is rated on a Likert scale ranging from 0 (Never) to 4 (Almost always) and indicates how often the caregiver has experienced the described situation. A total score ranging from 0 to 88 is calculated with increasing scores indicating greater burden experienced.
Change from baseline in the Zarit Caregiver Burden Interview (ZBI) total scores at a 3-week follow up period | The ZBI will be administered at baseline (i.e., prior to starting the study) and at a 3-week follow-up period.
  Caregiver burden will be assessed using the ZBI. The ZBI is a 22-item self-report questionnaire designed to measure the extent of the burden experienced by the caregivers in various dimensions (e.g., health, psychological well-being, finances, social) of their lives as a result of caregiving. Each item is rated on a Likert scale ranging from 0 (Never) to 4 (Almost always) and indicates how often the caregiver has experienced the described situation. A total score ranging from 0 to 88 is calculated with increasing scores indicating greater burden experienced.
Change from after the 2-week period in the Zarit Caregiver Burden Interview (ZBI) total scores at a 3-week follow up period | The ZBI will be administered after a 2-week period and at a 3-week follow-up period.
  Caregiver burden will be assessed using the ZBI. The ZBI is a 22-item self-report questionnaire designed to measure the extent of the burden experienced by the caregivers in various dimensions (e.g., health, psychological well-being, finances, social) of their lives as a result of caregiving. Each item is rated on a Likert scale ranging from 0 (Never) to 4 (Almost always) and indicates how often the caregiver has experienced the described situation. A total score ranging from 0 to 88 is calculated with increasing scores indicating greater burden experienced.
Change from baseline in the Perceived Stress Scale-10 (PSS-10) total scores at 2 weeks | The PSS-10 will be administered at baseline (i.e., prior to starting the study) and immediately after the end of the intervention period (i.e., after a 2-week period).
  Perceived stress over the course of the intervention will be assessed using the PSS-10. The PSS-10 is a 10-item self-report questionnaire designed to measure general feelings of stress and overload in the past four weeks. Each item is rated on a 5-point Likert scale ranging from 0 (Never) to 4 (Very often). A total score ranging from 0 to 40 is calculated with increasing scores indicating greater stress.
Change from baseline in the Perceived Stress Scale-10 (PSS-10) total scores at a 3-week follow up period | The PSS-10 will be administered at baseline (i.e., prior to starting the study) and at a 3-week follow-up period.
  Perceived stress over the course of the intervention will be assessed using the PSS-10. The PSS-10 is a 10-item self-report questionnaire designed to measure general feelings of stress and overload in the past four weeks. Each item is rated on a 5-point Likert scale ranging from 0 (Never) to 4 (Very often). A total score ranging from 0 to 40 is calculated with increasing scores indicating greater stress.
Change from after a 2-week period on the Perceived Stress Scale-10 (PSS-10) total scores at a 3-week follow up period | The PSS-10 will be administered after a 2-week period and at a 3-week follow-up period.
  Perceived stress over the course of the intervention will be assessed using the PSS-10. The PSS-10 is a 10-item self-report questionnaire designed to measure general feelings of stress and overload in the past four weeks. Each item is rated on a 5-point Likert scale ranging from 0 (Never) to 4 (Very often). A total score ranging from 0 to 40 is calculated with increasing scores indicating greater stress.
Change from baseline in the Short-Form Health Survey-12 (SF-12) scores at 2 weeks | The SF-12 will be administered at baseline (i.e., prior to starting the study) and immediately after the end of the intervention period (i.e., after a 2-week period).
  Overall well-being will be assessed using the SF-12. The SF-12 was derived from the original 30-item scale and is a self-report questionnaire that measures two dimensions of overall health: physical and mental. Accordingly, the scale consists of a Physical Component (SF-PC) and a Mental Component (SF-MC). Each item in the SF-12 is scored according to the scale's scoring algorithm and combined for each subscale. Total and subscale (SF-PC and SF-MC) scores range from 0 to 100, with increasing normed scores indicating better health and a score of 50 is average.
Change from baseline in the Short-Form Health Survey-12 (SF-12) scores at a 3-week follow up period | The SF-12 will be administered at baseline (i.e., prior to starting the study) and at a 3-week follow-up period.
  Overall well-being will be assessed using the SF-12. The SF-12 was derived from the original 30-item scale and is a self-report questionnaire that measures two dimensions of overall health: physical and mental. Accordingly, the scale consists of a Physical Component (SF-PC) and a Mental Component (SF-MC). Each item in the SF-12 is scored according to the scale's scoring algorithm and combined for each subscale. Total and subscale (SF-PC and SF-MC) scores range from 0 to 100, with increasing normed scores indicating better health and a score of 50 is average.
Change from after a 2-week period in the Short-Form Health Survey-12 (SF-12) scores at a 3-week follow up period | The SF-12 will be administered immediately after the end of the intervention period (i.e., after a 2-week period) and at a 3-week follow-up period.
  Overall well-being will be assessed using the SF-12. The SF-12 was derived from the original 30-item scale and is a self-report questionnaire that measures two dimensions of overall health: physical and mental. Accordingly, the scale consists of a Physical Component (SF-PC) and a Mental Component (SF-MC). Each item in the SF-12 is scored according to the scale's scoring algorithm and combined for each subscale. Total and subscale (SF-PC and SF-MC) scores range from 0 to 100, with increasing normed scores indicating better health and a score of 50 is average.
Change from baseline in the Dementia Knowledge Assessment Tool Version 2 (DKAT2) total scores at 2 weeks | The DKAT2 will be administered at baseline (i.e., prior to starting the study) and immediately after the end of the intervention period (i.e., after a 2-week period).
  Knowledge about dementia will be assessed using the DKAT2. DKAT2 is a 21-item self-report questionnaire designed to assess overall knowledge about dementia and dementia care among caregivers and health care staff. The DKAT2 expands from the previous DKAT version (i.e., DKAT1) by including items that are also be pertinent to family members and informal caregivers of people with dementia. Thirteen items in the scale are correct and eight items are incorrect. As such, reversal ratings are required and a score is calculated by summing the total number of correct responses ranging from 0 to 21, with higher scores indicating greater overall knowledge about dementia.
Change from baseline in the Dementia Knowledge Assessment Tool Version 2 (DKAT2) total scores at a 3-week follow up period | The DKAT2 will be administered at baseline (i.e., prior to starting the study) and at a 3-week follow-up period.
  Knowledge about dementia will be assessed using the DKAT2. DKAT2 is a 21-item self-report questionnaire designed to assess overall knowledge about dementia and dementia care among caregivers and health care staff. The DKAT2 expands from the previous DKAT version (i.e., DKAT1) by including items that are also be pertinent to family members and informal caregivers of people with dementia. Thirteen items in the scale are correct and eight items are incorrect. As such, reversal ratings are required and a score is calculated by summing the total number of correct responses ranging from 0 to 21, with higher scores indicating greater overall knowledge about dementia.
Change from after a 2-week period in the Dementia Knowledge Assessment Tool Version 2 (DKAT2) total scores at a 3-week follow up period | The DKAT2 will be administered immediately after the end of the intervention period (i.e., after a 2-week period) and at a 3-week follow-up period.
  Knowledge about dementia will be assessed using the DKAT2. DKAT2 is a 21-item self-report questionnaire designed to assess overall knowledge about dementia and dementia care among caregivers and health care staff. The DKAT2 expands from the previous DKAT version (i.e., DKAT1) by including items that are also be pertinent to family members and informal caregivers of people with dementia. Thirteen items in the scale are correct and eight items are incorrect. As such, reversal ratings are required and a score is calculated by summing the total number of correct responses ranging from 0 to 21, with higher scores indicating greater overall knowledge about dementia.

SECONDARY OUTCOMES:
Total System Usability Scale (SUS) score after the 2 week period | The SUS will be administered after the end of the intervention period (i.e., after a 2 week period) for app-using participants.
  Overall app usability will be assessed using the SUS. SUS is a 10-item self-report questionnaire designed to efficiently assess the usability of a technology or product. Each item is rated on a Likert scale ranging from 1 (Strongly disagree) to 5 (Strongly agree). An adjustment rating is needed to account for alternating positive and negative tone items in the instrument. Accordingly, 1 point is subtracted from the raw score of the odd-numbered items, while the raw score of even-numbered items is subtracted from 5. Next, the adjusted scores are added and multiplied by 2.5 to get the standard SUS score. A total score ranging from 5 to 100 is calculated with increasing scores indicating greater agreement and technology usability.
Total Mobile App Rating Scale Subjective App Quality score after the 2 week period | The MARS Subjective App Quality Rating will be administered after the end of the intervention period (i.e., after a 2-week period) for app-using participants.
  The subjective quality section of the MARS will be used to assess the user's overall app satisfaction. MARS is a 23-item questionnaire designed to assess the quality of mHealth applications. Each item is rated on a Likert scale ranging from 1 (inadequate) to 5 (excellent). The questionnaire includes a 4-item app quality section. A total score is obtained by summing the scores for each item and ranges from 1 to 20, with higher scores indicating greater user quality rating and satisfaction. The four items in the scale assess user's likeliness to recommend/pay for app, extent to which the app stimulates repeated use, and overall app satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Louise IR Castillo, BSc (Hons), Principal Investigator — University of Regina; Thomas Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Yes
All and non-identified numeric data will be made available to other researchers, following the publication of the results, upon reasonable request for a period of at least 7 years. Textual data from the interviews will not be shared to protect participant anonymity.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be made available to other researchers, following the publication of the results, upon reasonable request for a period of at least 7 years.
Access Criteria: Requests by researchers who wish to access the data can be directed to Thomas.Hadjistavropoulos@uregina.ca

REFERENCES:
- [Background] Toye C, Lester L, Popescu A, McInerney F, Andrews S, Robinson AL. Dementia Knowledge Assessment Tool Version Two: development of a tool to inform preparation for care planning and delivery in families and care staff. Dementia (London). 2014 Mar 1;13(2):248-56. doi: 10.1177/1471301212471960. Epub 2013 Jan 16. PMID 24339059
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Stoyanov SR, Hides L, Kavanagh DJ, Zelenko O, Tjondronegoro D, Mani M. Mobile app rating scale: a new tool for assessing the quality of health mobile apps. JMIR Mhealth Uhealth. 2015 Mar 11;3(1):e27. doi: 10.2196/mhealth.3422. PMID 25760773
- [Background] Riffin C, Van Ness PH, Wolff JL, Fried T. Family and Other Unpaid Caregivers and Older Adults with and without Dementia and Disability. J Am Geriatr Soc. 2017 Aug;65(8):1821-1828. doi: 10.1111/jgs.14910. Epub 2017 Apr 20. PMID 28426910
- [Background] Brown EL, Ruggiano N, Li J, Clarke PJ, Kay ES, Hristidis V. Smartphone-Based Health Technologies for Dementia Care: Opportunities, Challenges, and Current Practices. J Appl Gerontol. 2019 Jan;38(1):73-91. doi: 10.1177/0733464817723088. Epub 2017 Aug 4. PMID 28774215
- [Background] Wozney L, Freitas de Souza LM, Kervin E, Queluz F, McGrath PJ, Keefe J. Commercially Available Mobile Apps for Caregivers of People With Alzheimer Disease or Other Related Dementias: Systematic Search. JMIR Aging. 2018 Dec 7;1(2):e12274. doi: 10.2196/12274. PMID 31518255
- [Background] Brooke, J. (1996). SUS-A quick and dirty usability scale. Usability evaluation in industry, 189(194), 4-7.
- [Background] Zarit, S., Orr, N. K., & Zarit, J. M. (1985). The hidden victims of Alzheimer's disease: Families under stress. NYU press.
- [Background] Seng BK, Luo N, Ng WY, Lim J, Chionh HL, Goh J, Yap P. Validity and reliability of the Zarit Burden Interview in assessing caregiving burden. Ann Acad Med Singap. 2010 Oct;39(10):758-63. PMID 21063635
- [Background] Bangor, A., Kortum, P. T., & Miller, J. T. (2008). An empirical evaluation of the system usability scale. Intl. Journal of Human-Computer Interaction, 24(6), 574-594.
- See also: CLEAR Dementia Care mobile app — https://play.google.com/store/apps/details?id=com.nhsct.clearcare